CLINICAL TRIAL: NCT03328182
Title: Assessment of AnchorFast Guard Subglottic ET (Endotracheal) Tube
Brief Title: Assessment of an Oral Endotracheal Subglottic Tube Holder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5855-I
Record Dates: First submitted 2017-10-16; First posted 2017-11-01 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- New oral endotracheal tube holder (Experimental): Single Study Product Arm
  Interventions: Device: New oral endotracheal tube holder

INTERVENTIONS:
Device: New oral endotracheal tube holder — The single arm study product is designed to hold a standard or subglottic ET tube.

SUMMARY:
This study is designed to assess the acceptability and usability of a new Endotracheal Tube (ET) holding device for an orally intubated patient.

DETAILED DESCRIPTION:
This is a multiple site prospective assessment of the study product in ICU settings. The study is comprised of each intubated subject wearing one study product until the device either needs to be changed or is no longer required by the subject. The study product is designed to hold a standard or subglottic ET tube and help reduce the potential for occlusion (blockage) of the tube.

ELIGIBILITY:
INCLUSION CRITERIA

1. Is 18 years of age or older and require oral tracheal intubation with subglottic ET tube size 6.0-8.0mm
2. Requires the use of a bite block per the hospital's standard of care
3. Has intact skin on and around application site, including cheeks and lips
4. Oral cavity is free of open sores, ulcers, wounds, and lesions
5. Subject or Legal Authorized representative (LAR) able to provide informed consent for the study
6. Is qualified to participate in the opinion of the Investigator, or designee

EXCLUSION CRITERIA

1. Has actual or perceived loose teeth, is without teeth, or is unable to wear upper dentures
2. Has facial hair that interferes with the adhesion of the skin barrier pads
3. Has a clinically significant skin disease or condition, or damaged skin on the application site, such as psoriasis, eczema, atopic dermatitis, active cancer, sores, sunburns, scars, moles
4. Has a medical condition, surgery or a procedure that prevents the proper application of the device, including placement of the neck strap.
5. Has a known or stated allergy to adhesives
6. Currently is participating in any clinical study which may affect the performance of the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vander Werff, MD, Principal Investigator — Legacy Mount Hood Medical Center; Brian Young, MD, Principal Investigator — 1. Legacy Emanuel Hospital & Health Center 2. Legacy Good Samaritan Medical Center; Arash Afshinnik, MD, Principal Investigator — Community Regional Medical Center
Locations (4):
- United States (4):
  - Community Regional Medical Center, Fresno, California
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital & Health Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buckley JC, Brown AP, Shin JS, Rogers KM, Hoftman NN. A Comparison of the Haider Tube-Guard(R) Endotracheal Tube Holder Versus Adhesive Tape to Determine if This Novel Device Can Reduce Endotracheal Tube Movement and Prevent Unplanned Extubation. Anesth Analg. 2016 May;122(5):1439-43. doi: 10.1213/ANE.0000000000001222. PMID 26983051
- [Background] Mohammed, H & Hassan, M. (2015). Endotracheal tube securements: Effectiveness of three techniques among orally intubated patients. Egyptian Journal of Chest Diseases and Tuberculosis 64:183-196

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Oral Endotracheal Tube Holder
Started | 34
Completed | 30
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2
Not completed — No Product Evaluated | 1

BASELINE CHARACTERISTICS:
Population: Enrolled patients found eligible per Inclusion/Exclusion Criteria
Arm/Group | New Oral Endotracheal Tube Holder
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 52.5 [21 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Acceptability With Study Product
Description: The overall acceptability relating to general experience with the study product during use will be rated with a 5-point Likert scale ranging from 1=Very Unacceptable to 5=Very Acceptable
Time Frame: At product removal (maximum 29 days of patient wearing product)
Measure: Count of Participants; unit: Participants
Arm/Group | New Oral Endotracheal Tube Holder
Number analyzed (Participants) | 30
Participants
  Very Acceptable | 13
  Acceptable | 15
  Neither acceptable nor acceptable | 0
  Unacceptable | 2
  Very Unacceptable | 0

2. Primary Outcome: Usability of Study Product
Description: The usability of the study product at application and at removal.
Time Frame: At application and product removal (maximum 29 days of patient wearing product)
Measure: Count of Participants; unit: Participants
Arm/Group | New Oral Endotracheal Tube Holder
Number analyzed (Participants) | 30
Participants
  Ease of application: Very easy to apply | 20
  Ease of application: Easy to apply | 8
  Ease of application: Neither easy nor difficult to apply | 1
  Ease of application: Difficult to apply | 1
  Ease of application: Very difficult to apply | 0
  Ease of application: Not Applicable | 0
  Ease of removal: Very easy to apply | 18
  Ease of removal: Easy to apply | 7
  Ease of removal: Neither easy nor difficult to apply | 2
  Ease of removal: Difficult to apply | 1
  Ease of removal: Very difficult to apply | 0
  Ease of removal: Not Applicable | 2

ADVERSE EVENTS:
Time Frame: maximum 29 days of patient wearing product
Description: Adverse Events were determined via standardized study investigator assessment forms. All Adverse Events are reported irrespective of relation to study product.
Arm/Group | New Oral Endotracheal Tube Holder
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Oral Endotracheal Tube Holder (N=30)
Death (Infections and infestations) | 1 (1) — Patient passed due to sepsis progression--not related to device
Oral Bleeding (General disorders) | 1 (1) — Patient constantly was biting for over 24 hours after product placement before oral bleeding occurred. Oral bleeding was exacerbated significantly by the heparin drip and other anticoagulation he was on while in the ICU.
Loose teeth (General disorders) | 1 (1) — Loose teeth due to prolonged biting, probably NOT related to study device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Oral Endotracheal Tube Holder (N=30)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) — Skin lesion on patient's skin, below nose, but above upper outer lip. Lesion could be due to a herpetic lesion or an underlying skin condition not previously identified/documented. Investigator indicated AE was probably not related to study device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 18 months from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT03328182/Prot_SAP_000.pdf